CLINICAL TRIAL: NCT03018379
Title: Assessment Study of Body Composition, Energy Expenditure and Physical Activity to Inform Design and Improve Interventions for the Prevention and Control of Obesity and Related Health Risks Among Schoolchildren and Adolescent Aged 8 to 14 Years in Morocco
Brief Title: Body Composition, Dietary Behaviors, Energy Expenditure and Physical Activity Among Moroccan Schoolchildren and Adolescents
Status: Completed | Type: Observational
Sponsor: Centre National De L'énergie, Des Sciences Et Techniques Nucléaires (Other Government)
Collaborators: Ministry of National Education, Morocco (Other Government); Ibn Tofail University, Morocco (Unknown); International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Asmaa El Hamdouchi, Principal Investigator, Centre National De L'énergie, Des Sciences Et Techniques Nucléaires
Other Study IDs: RAF642
Record Dates: First submitted 2016-12-23; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Body Composition; Physical Activity
Keywords: Obesity; Body composition; energy expenditure; sedentarity; dietary behaviors
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Assessment of body composition: The collection of the samples and the analyses were undertaken according to the guidelines of the International Atomic Energy Agency. In brief, after having emptied the bladder, each participant provided a predose saliva sample using a cotton ball.A 99.8 % deuterium dose of 0.5 g per kg body weight was given orally to the participant. The postdose sample was collected from 3h to 4h after the administration of the dose. The saliva samples were stored at 20°C until analysis by Fourier transform infrared spectroscopy (FTIR).
- Assessment of energy expenditure: Each participant provided a predose urine sample. A dose of doubly labelled water 2.625 ml per kg body weight was given orally to the participant.
  The post dose sample was collected at 3h to 4h , and on days 3, 7 and 14 after dosing. An aliquot of those samples were stored at 20°C in tightly sealed containers until analysis by isotope-ratio mass spectrometry (IRMS).
- Assessment of physical activity: The participants were instructed to wear the accelerometer triaxial (GT3X+) attached to an elasticized belt around the waist, once they woke up until bed time at night for 7 consecutive days and to remove the accelerometer any time they were to perform activities that involve the use of water and when going to bed.

SUMMARY:
Considering the increasing public health concern the obesity in Morocco, the aim of the present study was to use isotope techniques to assess body fat, total energy expenditure and physical activity to inform design and improve interventions for the prevention and control of obesity and related health risks such as diabetes and elevated blood pressure among children and adolescents. Specific objectives of the trial: 1. Determine the extent of obesity and physical activity levels in children and adolescents to design effective interventions in the school setting. 2.Propose alternative field based techniques for assessing body composition and physical activity that could be used in largescale situation assessments and in assessing interventions to address obesity and risk related health care. * For body composition: BMI z-score, waist circumference, waist measurement at height. * For physical activity: Questionnaire, Accelerometers 3. To identify factors contributing to the development of obesity and related health risks in schoolchildren and adolescents. 4. Collaborate with stakeholders (government, schools and / or colleges, communities and development partners) in designing interventions to address obesity and health risks. 5. To recommend to stakeholders the most effective interventions in schools to prevent and combat obesity and health risks in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Aged between 8 to 14 years old

Exclusion Criteria:

* Hypo or hypervolemic conditions including diet
* Diuretics and oedema
* Private schools
* Rural area

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Moroccan children and adolescents recruited from public urban schools.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Assessment of body composition using deuterium dilution technique | 1 year
  Each participant provided a predose saliva sample. The postdose sample was collected from 3h to 4h after the administration of the dose.
Assessment of energy expenditure using isotopes dilution techniques | 1 year
  Each participant provided a predose urine sample. The postdose urine samples were collected after 3h to 4h and on days 3, 7 and 14.
Assessment of physical activity levels using accelerometry triaxial (GT3X+) | 2 years 6 months

SECONDARY OUTCOMES:
Assessment of dietary intake using 24h recall questionnaire | 6 months
Assessment of physical activity levels using physical activity questionnaire for children (PAQ-C) | 2 years 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa EL HAMDOUCHI, Dr, Principal Investigator — Unité Mixte de Recherche en Nutrition, CNESTENIbn Tofail university